CLINICAL TRIAL: NCT03043235
Title: Race Adiposity Interactions Regulate Mechanisms Determining Insulin Sensitivity
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Barbara Gower, Prinicipal Investigator, University of Alabama at Birmingham
Other Study IDs: 2237
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Insulin Sensitivity; Fat; Liver
MeSH Terms: conditions — Insulin Resistance; Fatty Liver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be used to identify ancestry. This information is needed to understand why African Americans and Caucasians have different risks for developing certain diseases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- African American Females: No intervention
- African American Males: No intervention
- Caucasian Females: No intervention
- Caucasian Males: No intervention

SUMMARY:
This research study will examine how ethnic/racial background, body composition (%body fat), and the location of body fat affect the ability of the hormone insulin to promote uptake of blood sugar in persons who are 19 to 45 years of age. When insulin is ineffective in promoting blood sugar uptake, this condition is termed "insulin resistance." Insulin resistance plays a major role in the development of chronic metabolic diseases (such as type 2 diabetes, cardiovascular disease, and cancer), many of which differ with race. Previous studies suggest that insulin resistance is higher in African-Americans (AA) vs. European-Americans (EA). However, results from these studies remain unclear due to different testing measures used for insulin resistance as well as differences in body fat between individuals. Results from this research study may help explain why insulin resistance differs with genetic background and may guide development of personalized treatment strategies with implications for several chronic metabolic diseases (e.g., type 2 diabetes, cardiovascular disease, and cancer).

DETAILED DESCRIPTION:
Insulin resistance plays a major role in the etiology of chronic metabolic diseases, many of which differ with race/ethnicity. Previous studies using mainly indirect methods suggest that insulin sensitivity is lower in AA vs. EA. Our preliminary data using the reference standard glucose clamp indicate that in lean individuals, insulin sensitivity is lower among AA, while in obese individuals, insulin sensitivity is higher among AA. We hypothesize that this race/body mass index (BMI) interaction may be explained in part by significantly lower visceral and hepatic fat accumulation in AA. Conversely, based on our preliminary data, we hypothesize that inherently greater oxidative stress impairs insulin sensitivity even in AA, explaining lower insulin sensitivity in lean AA vs. EA. We propose to test these hypotheses by prospectively comparing skeletal muscle and hepatic insulin sensitivity in healthy lean, overweight, and obese AA and EA using the hyperinsulinemic isoglycemic glucose clamp. Analysis of ancestral genes will permit simultaneous assessment of the contribution of ancestry to main outcomes.

ELIGIBILITY:
Inclusion Criteria:

* African American or Caucasian
* Body Mass Index 19-45
* Do NOT have diabetes
* Exercise less than 2 hours per week
* Are willing to travel to UAB for 2 screens and 4 testing visits

Exclusion Criteria:

* Diabetes
* Any major medical conditions or medications that interfere with study outcomes

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: African American and Caucasian Males and Females between 19-45 years old
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2014-01-08 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Hyperinsulinemic isoglycemic glucose clamp | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gower, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fisher G, Tay J, Warren JL, Garvey WT, Yarar-Fisher C, Gower BA. Sex and race contribute to variation in mitochondrial function and insulin sensitivity. Physiol Rep. 2021 Oct;9(19):e15049. doi: 10.14814/phy2.15049. PMID 34605220